CLINICAL TRIAL: NCT07344623
Title: Factors Associated With Clinical Pregnancy Outcomes in Intrauterine Insemination (IUI) Cycles
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2025.831
Record Dates: First submitted 2025-12-30; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Reproductive Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypotheses:

We hypothesize that variations in hormonal profiles (LH, estradiol, progesterone) during ovarian stimulation, follicular response, endometrial characteristics, and sperm quality parameters are significantly associated with clinical pregnancy outcomes in intrauterine insemination (IUI) cycles.

Aims

* To investigate the association between hormonal profiles on the trigger day (LH, estradiol, progesterone), follicular response, endometrial thickness, and sperm parameters with clinical pregnancy outcomes in IUI cycles.
* To develop and validate a predictive model for clinical pregnancy incorporating key determinants such as female age, hormonal response, endometrial characteristics, and sperm quality.
* To compare natural and gonadotropin-stimulated IUI cycles in terms of hormonal profiles, pregnancy outcomes, and cost-effectiveness.

Primary Outcome Clinical pregnancy rate (CPR), defined as the presence of a gestational sac with a fetal heartbeat on ultrasound at approximately 6 weeks of gestation following intrauterine insemination.

Secondary Outcomes

* Biochemical pregnancy rate.
* Ongoing pregnancy rate
* Live birth rate

DETAILED DESCRIPTION:
Statistical Analysis

Each sub-study will employ specific analytical approaches:

* Univariate and multivariate logistic regression for associations
* Mediation and interaction analysis
* ROC and AUC analysis for predictive modeling
* Machine learning for model development
* Cost-effectiveness evaluated via incremental cost per clinical pregnancy

Consent

This is a retrospective study, and thus, there is no need for a written informed consent.

Sample Size All eligible IUI cycles, estimated to be approximately 3000 cycles, will be included

ELIGIBILITY:
Inclusion Criteria:

* Couples who underwent at least one IUI-intrauterine insemination cycle.

Exclusion Criteria:

* Couples who used donor sperm.
* Cases with missing core outcome data

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This retrospective study will include all infertile couples who underwent intrauterine insemination (IUI) at the Asisted Reproductive Unit, Department of Obstetrics and Gynaecology, Prince of Wales Hospital, Hong Kong, China
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate (CPR) | 6 weeks gestation and ultrasound scanning will be performed to confirm at least one gestational sac around 2 to 3 months after IUI.
  Rate of clinical pregnancy outcome in subjects undergoing IUI

SECONDARY OUTCOMES:
Biochemical pregnancy rate | Up to 12 weeks
  Rate of biochemical pregnancy outcome in subjects undergoing IUI
Ongoing pregnancy rate | Up to 12 weeks
  Rate of Ongoing pregnancy outcome in subjects undergoing IUI
live birth rate | Up to 40 weeks
  Rate of live birth rate outcome in subjects undergoing IUI

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided